CLINICAL TRIAL: NCT01142661
Title: Compassionate Use of Eribulin for the Treatment of Advanced Breast Cancer Refractory to All Other Marketed Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-399
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer refractory to all commercially available therapies
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eribulin mesylate (Experimental)
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin Mesylate: A dose of 1.4 mg/m^2 given intravenously on Day 1 and Day 8 of a 21 day cycle, continued until disease progression, unacceptable toxicity or death.

SUMMARY:
The purpose of this study is to provide eribulin to patients with advanced breast cancer who have no other treatment options and therapy is requested by an Investigator.

DETAILED DESCRIPTION:
This compassionate use program will consist of a Pretreatment Phase and a Treatment Phase. Patients with locally advanced or metastatic breast cancer who fulfill the eligibility criteria may be treated. Safety data will be collected, but a minimal amount of other data will also be collected.

ELIGIBILITY:
Inclusion Criteria

In order to receive eribulin under this protocol, the subjects oncologist must have documented experience treating subjects with eribulin in a prior clinical study. Subjects who meet all of the following criteria will be included in the treatment protocol:

1. Recurrent, locally advanced or metastatic breast cancer that has progressed on or after the last anti-cancer therapy.
2. Prior treatment with, ineligibility for, or commercial unavailability of each of the following therapies:

   * Anthracyclines, taxanes, and capecitabine.
   * Ixabepilone in countries where this agent is marketed.
   * Trastuzumab for Her-2 positive disease.
   * Hormonal therapy in hormone receptor-positive disease.
   * All other marketed therapies, eg, gemcitabine or vinorelbine, used for the treatment of advanced breast cancer.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
4. Serum creatinine </= 2.0 mg/dL or creatinine clearance >/= 40 mL/min according to Cockcroft and Gault formula.
5. Absolute neutrophil count >/= 1.5 x 10^9/L, hemoglobin >/= 10 g/dL (can be corrected by growth factor or transfusion), and platelet count >/= 100 x 10^9/L.
6. Total bilirubin </= 1.5 x upper limit of normal (ULN). Alkaline phosphatase (AP), alanine aminotransferase, and aspartate aminotransferase </= 3 x ULN (</= 5 x ULN in case of liver metastases). In case AP is >3 x ULN (in absence of liver metastases) or >5 x ULN (in presence of liver metastases) AND subject also is known to have bone metastases, the liver specific AP must be separated from the total and used to assess the liver function instead of the total AP.
7. Are willing and able to comply with all aspects of the treatment protocol.
8. Provide written informed consent.
9. Females, age >/= 18 years.
10. Female subjects of childbearing potential must agree to be abstinent or to use a highly effective methods of contraception (eg, condom + spermicide, condom + diaphragm with spermicide, intra-uterine device, or have a vasectomised partner) having started for at least one menstrual cycle prior to starting eribulin and throughout the entire treatment period and for 30 days (longer if appropriate) after the last dose of eribulin. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria Subjects who meet any of the following criteria will be excluded from participation in the treatment protocol:

1. Eligible for any other eribulin study that is open in the same region.
2. Existing anti-cancer therapy-related toxicities of Grade >/= 2, except that alopecia and Grade 2 neuropathy are acceptable.
3. History of congestive heart failure with New York Heart Association Classification >II, unstable angina, myocardial infarction within the past 6 months, serious cardiac arrhythmia.
4. Electrocardiogram with QTc interval >/= 500 msec based upon Bazett's formula (QTcB).
5. The Investigator believes the subject to be medically unfit to receive eribulin or unsuitable for any other reason.
6. Females who are pregnant (positive B-hCG test) or breastfeeding.
7. Subject with hypersensitivity to eribulin or any of the excipients.
8. Subjects with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this treatment protocol. Any signs (eg, radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks before starting the treatment protocol.
9. Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the subject's ability to safely complete the treatment protocol.
10. Subjects who are known to be human immunodeficiency virus positive because the neutropenia caused by the eribulin treatment may make such subjects particularly susceptible to infection.
11. Subjects with meningeal carcinomatosis.
12. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
13. Subjects who have received any of the following treatments within the specified period before the start of treatment:

    * Any investigational drug, chemotherapy, radiation, or biological or targeted therapy within 2 weeks.
    * Hormonal therapy within 1 week.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (5):
- United States (5):
  - La Verne, California
  - Nyack, New York
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 5 centers in the US during the period of Aug 2010 to Aug 2011.
Groups:
- Eribulin Mesylate: Eribulin Mesylate : Eribulin Mesylate: A dose of 1.4 mg/m^2 given intravenously on Day 1 and Day 8 of a 21 day cycle, continued until disease progression, unacceptable toxicity or death.
Period: Overall Study
Arm/Group | Eribulin Mesylate
Started | 9
Completed | 5
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: General safety will be assessed by monitoring and recording the number of patients with adverse events (serious and nonserious) for duration of treatment which continued until disease progression, unacceptable toxicity or death.
Time Frame: For duration of treatment, an average of 5 months
Measure: Number; unit: participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
participants | 9

2. Primary Outcome: Safety
Description: General safety will be assessed by monitoring and recording the number of patients with serious adverse events for duration of treatment which continued until disease progression, unacceptable toxicity or death.
Time Frame: For duration of treatment, an average of 5 months
Measure: Number; unit: participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
participants | 7

ADVERSE EVENTS:
Arm/Group | Eribulin Mesylate
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=9)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Alcohol Poisoning (Musculoskeletal and connective tissue disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=9)
Neutropenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Congenital, familial and genetic disorders) | 1
Tachyarrhythmia (Eye disorders) | 1
Lacrimation Increased (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision Blurred (Gastrointestinal disorders) | 1
Vision Impairment (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Hernia (General disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 1
Mouth Ulceration (Investigations) | 1
Oral Discomfort (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Peripheral Edema (General disorders) | 2
Cyst (General disorders) | 1
Mucosal Inflammation (General disorders) | 1
Oral Herpes (Infections and infestations) | 1
Skin Infection (Injury, poisoning and procedural complications) | 1
Urinary Tract Infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Neutrophil Count Decreased (Investigations) | 2
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
Hemoglobin Decreased (Investigations) | 1
Occult Blood Positive (Investigations) | 1
Decreased Appetite (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fluid Retention (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Pregnancy, puerperium and perinatal conditions) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Upper Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Insomnia (Psychiatric disorders) | 1
Phlebitis (Vascular disorders) | 1
Phlebitis Superficial (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No